CLINICAL TRIAL: NCT02675842
Title: Investigation of Cannabis for Pain and Inflammation in Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: funding
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Diana Martinez, Associate Professor of Psychiatry at CUMC, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7221
Record Dates: First submitted 2016-01-28; First posted 2016-02-05 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Smoked Cannabis High CBD/low THC (Active Comparator): Participants will visit the research laboratory 3-5 days a week over 6 weeks to be administered 1-2 Cannabis cigarettes (15.76% CBD; 3.11% -9-THC) over the course of 2-3 hours.
  Interventions: Drug: Smoked Cannabis High CBD/low THC
- Smoked Placebo Cannabis Low CBD/low THC (Placebo Comparator): Participants will visit the research laboratory 3-5 days a week over 6 weeks to be administered 1-2 Cannabis cigarettes Cannabis (0.0% CBD/ 0.01% -9-THC) over the course of 2-3 hours.
  Interventions: Drug: Smoked Placebo Cannabis Low CBD/low THC

INTERVENTIONS:
Drug: Smoked Cannabis High CBD/low THC — Participants will visit the research laboratory 3-5 days a week over 6 weeks to be administered 1-2 Cannabis cigarettes (15.76% CBD; 3.11% -9-THC) over the course of 2-3 hours.
  Arms: Smoked Cannabis High CBD/low THC
Drug: Smoked Placebo Cannabis Low CBD/low THC — Participants will visit the research laboratory 3-5 days a week over 6 weeks to be administered 1-2 Cannabis cigarettes Cannabis (0.0% CBD/ 0.01% -9-THC) over the course of 2-3 hours.
  Arms: Smoked Placebo Cannabis Low CBD/low THC

SUMMARY:
Radiation therapy to the chest is used in late stage lung cancer, and it often leads to inflammation of the esophagus. The inflammation is expected to occur in about 75% of patient, and usually begin within a week of starting radiation therapy. The esophagitis causes pain and difficulty eating. It can also result in stopping or delaying treatment.Radiation therapy to the chest is used in late stage lung cancer, and it often leads to inflammation of the esophagus. The inflammation is expected to occur in about 75% of patient, and usually begin within a week of starting radiation therapy. The esophagitis causes pain and difficulty eating. The endocannabinoid system is prominent in the gastrointestinal system, and cannabis has been shown to greatly inhibit inflammation. The compound (-)-trans-Δ9-tetrahydrocannabinol (Δ-9-THC) has effects that reduce inflammation and pain. Cannabidiol is a component of cannabis that does not produce subjective or intoxicating effects, but also has prominent anti-inflammatory properties.

The goal of this study is to perform a double-blind, placebo-controlled study to investigate the efficacy of cannabis, compared to placebo, in participants undergoing RT (Radiation Therapy) for lung cancer. Cannabis that has a high concentration of cannabidiol will be used , which is a cannabinoid that does not change perception or produce intoxication, and low in Δ-9-THC. In this way, the hope is to maximize the benefit of cannabis, while lowering the possible side effects of cannabis in medically ill participants.

DETAILED DESCRIPTION:
Study Outline

Patients will be referred to the study from their physician, who will have the patients medically cleared for participation.

The patients will then undergo additional screening for the study. A study physician will review all study procedures with potential participants, including the potential side effects. Patients will be shown the facilities and informed of being monitored at all times.

Patients will be randomized using a randomization and assigned to one of two groups: cannabis (15.76% CBD; 3.11% Δ-9 -THC) vs "placebo" cannabis (0.0% CBD/ 0.01% Δ-9-THC).

Participants will visit the Marijuana Research Laboratory, 3-5 days a week over 6 weeks to be administered 1-2 cannabis cigarettes over the course of a 2-3 hour session. Two cannabis conditions will be tested: Placebo (0.01% THC; 0.00% CBD) and CBD:THC (15.76% CBD; 3.11% THC) provided by the National Institute on Drug Abuse.

Participants will undergo baseline measurements of mood, and physical symptoms and will then be given 2 NIDA (National Institute on Drug Abuse) cannabis cigarettes, which can be consumed as smoking or with a vaporizer in a ventilated room. After the 90 minutes of cannabis availability end, participants will be asked to remain in the laboratory for an additional 45 minutes to allow the effects of the cannabis to wear off.

Participants will undergo baseline measurements of mood, and physical symptoms and will then be given the equivalent of 2 NIDA cannabis cigarettes. Cardiovascular and subjective effects measures of mood, abuse liability and drug tolerability will be collected at baseline, at the end of the 90 minutes of cannabis availability and at the end of the session. Detailed measures of food intake (caloric content, macronutrient intake) will be recorded beginning immediately after cannabis administration and for the duration of the session. In addition to visual analog scales, participants will be asked to complete measures of mood and cannabis effects at screening, before, during and after the session. Participants will be assessed at the end of the session by an experienced clinician.

Opioid use: Participants will be asked to provide the number of opioid medications taken as follows: 1) at baseline (in the week prior to starting sessions); and 2) at each session, participants will be asked about opioid use since the previous session. The amount of opioids used will be converted to oral morphine equivalents and tallied for each day.

Food intake: Participants will be asked to complete a daily food diary for the duration of the study. Detailed measures of food intake (caloric content, macronutrient intake) will also be recorded during the cannabis sessions. Participants will also be weighed weekly.

PET (Positron Emission Tomography) scans: As part of their clinical care, patients receive a PET/CT scan using the radiotracer [18F]FDG with a low dose CT for attenuation correction and anatomic localization. This data will be requested from the PET center, with the participants consent, in order to assess the extent of esophagitis in the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Lung Cancer receiving RT.
2. Age 21- 60
3. Able to give informed consent, and comply with study procedures.
4. History of previous experience with smoking or marijuana. On PFTs (Pulmonary Function Tests), participants must have an FEV1 (Forced Expiratory Volume in 1 second) of ≥ 1.2 liters/second or ≥ 50% predicted using the CDC reference value calculator.

Exclusion Criteria:

1. Meet DSM-V criteria for current major psychiatric illness, such as bipolar disorder, major depression, active suicidal intent, or psychosis, that could be exacerbated by the administration of cannabis.
2. Meet criteria for major neurological disorder, such as mild cognitive impairment or neurodegenerative disorders (such as movement disorders, dementia), that could be exacerbated by the administration of cannabis.
3. Women who are not practicing an effective form of birth control (condoms, diaphragm, birth control pill, IUD) or currently pregnant
4. Current (weekly) use of cannabis.
5. Participants on supplemental oxygen
6. Participants with a history of substance use disorder other than nicotine, such as opiate disorder

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Change in pain ratings using The McGill Pain Questionnaire | 6 weeks
  Participants will be asked to rate their pain over the 6 weeks of receiving active cannabis vs placebo.
Change in sickness-related impairment using the Sickness Impact Profile Questionnaire | 6 weeks
  Participants will be asked to rate physical symptoms for the 6 weeks of the study.
changes in physical and emotional well being using RAND 36 item medical outcomes survey | 6 weeks
Changes in symptoms of pain using 9 item Brief Pain Inventory | 6 weeks
Changes in quality of life using the Multidimensional Index of Life Quality (MILQ) Questionnaire | 6 weeks
changes in symptoms of pain, tiredness and well-being using the Edmonton Symptom | 6 weeks
Change in symptoms of pain, mood and appetite using the System (ESAS) Questionnaire | 6 weeks

SECONDARY OUTCOMES:
Assessment of subjective effects using VAS | 6 weeks
  The visual analog scales (VAS) will be used to investigate the subjective effects while participants are in the laboratory.
change in eating measured using food diary | weekly for 6 weeks
  Participants will be asked to complete a food diary during the 6 weeks and will be weighed weekly during the study.
Change in mood using the Hamilton Depression Rating Scale | 6 weeks
  Hamilton Depression Rating Scale will be used to assess mood during the 6 weeks of the study.
Change in mood Hamilton Anxiety Rating Scale | 6 weeks
  Hamilton Anxiety Rating Scale will be used to assess mood during the 6 weeks of the study.
Change in mood using the Montgomery-Asberg Depression Rating Scale | 6 weeks
  The Montgomery-Asberg Depression Rating Scale will be used to assess the participants' mood throughout the six weeks of the study.
Change in mood and quality of life using the Columbia Suicide Severity Rating Scale | 6 weeks
change in cognitive status using the Short Portable Mental Status Questionnaire (SPMSQ) | 6 weeks
Change in symptom prevalence using the Memorial Symptom Assessment Scale (MSAS) | 6 weeks
Change in physiological state using the Mental Health Inventory-5 (MHI-5) Questionnaire | 6 weeks
Change in opioid use using the Opioid use Questionnaire | Daily for 6 weeks
  Participants will be asked to provide to the number of opioid medications taken. The amount of opioids used will be converted to oral morphine equivalents and tallied for each day.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Martinez, MD, Principal Investigator — Columbia University/NYSPI

IPD SHARING:
Plan to Share IPD: No